CLINICAL TRIAL: NCT07029152
Title: Screening for Anal Cancer in MSM Using PrEP
Brief Title: Screening for Anal Cancer in Men Who Have Sex With Men Using Pre-Exposure Prophylaxis
Acronym: SCOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: A.M.L. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SCOPE
Record Dates: First submitted 2025-06-02; First posted 2025-06-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Anal Cancer; Squamous Intraepithelial Lesions; HSIL, High Grade Squamous Intraepithelial Lesions; LSIL, Low-Grade Squamous Intraepithelial Lesions; HPV; Squamous Cell Carcinoma
Keywords: HIV prevention; men who have sex with men; pre-exposure prophylaxis (PrEP); anal cancer
MeSH Terms: conditions — Anus Neoplasms; Squamous Intraepithelial Lesions; Carcinoma, Squamous Cell; Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSM group (Experimental): The MSM group consists of men who have sex with men (MSM) who are using Pre-Exposure Prophylaxis (PrEP) for HIV prevention.
  Participants in this group will undergo the following interventions:
  * Health and Quality of Life Questionnaires
  * Anal Smear Collection
  * High-Resolution Anoscopy (HRA)
  Interventions: Diagnostic Test: Anal smear; Behavioral: Self-administered questionnaire; Behavioral: EQ-5D-5L questionnaire; Diagnostic Test: High Resolution Anoscopy (HRA)

INTERVENTIONS:
Diagnostic Test: Anal smear — The intervention in this study involves the anal smear collection using the FLOQSwab® (COPAN, pouch type 502CS01). The swab is inserted 3-5 cm into the anal canal, reaching the transitional zone, the pressed against the canal wall and withdrawn in a spiral motion over approximately 20 seconds. After collection, the swab is immediately placed into a ThinPrep vial containing 20 ml of PreservCyt® and rinsed vigorously.
  The procedure is performed by a physician or trained study team member and is designed to be quick, minimally invasive, and comfortable for participants. The FLOQSwab®'s patient-friendly design reduces irritation and false-positive results in comparison to earlier methods.
  Samples collected in the ThinPrep PreservCyt® solution should be stored at room temperature and transferred to AML within a maximum of six weeks
Behavioral: Self-administered questionnaire — It includes questions related to:
  Socio-demographic characteristics Health-related issues Past HPV vaccination (indication? age at vaccination?) History of condylomata and/or other STIs Drug use, tobacco use, alcohol use Anal symptoms: discomfort, itch, pain, nodules, blood loss/discharge, constipation Sexual behavior Insertive/receptive intercourse, chemsex, number of sex partners (stable, occasional, anonymous), condom use.
Behavioral: EQ-5D-5L questionnaire — This questionnaire will be used after a negative HRA or during the communication of the results (per telephone) and during the treatment if indicated. This questionnaire assesses the impact of health conditions and treatments on person's quality of life. We will use an adapted version of the EQ-5D-5L. This modified version includes additional questions tailored to assess specific domains highlighted in the A-HRSI.
  The additional items cover:
  * Physical Symptoms: Question on anal symptoms such as pain, discharge, and burning sensations.
  * Impact on Physical Functioning: Question on how these symptoms affect daily activities, including work, sitting, and social interactions.
  * Impact on Psychological Functioning: Question on psychological and sexual well-being, including enjoyment and desire for sex, as well as challenges with intimacy.
Diagnostic Test: High Resolution Anoscopy (HRA) — HRA will be conducted using advanced tools, such as the Zeiss Extaro at UZ Brussel.
  HRA will be conducted at participating centers with expertise in the technique, including UZ Brussel, UZ Gent, UZ Leuven, UZ Antwerpen, CHU St Pierre, AZ Sint-Jan Brugge, and Citadelle Liège. However, all biopsy specimens will be sent to AML Lab for analysis and stored in the biobank (BB190002).
  In certain centers, HRA is performed using high-resolution scopes.

SUMMARY:
This study aims to learn more about anal cancer risk in men who have sex with men (MSM) who are using Pre-Exposure Prophylaxis (PrEP) to prevent HIV. Specifically, we want to check how common High-Grade Squamous Intraepithelial Lesions (HSIL) are in this group, how well anal swabs can screen for these lesions, and how having HSIL affects their quality of life. We'll also test if DNA methylation testing can give us extra information about the lesions.

The main questions the study aims to answer are:

* How common are HSIL in MSM using PrEP?
* How accurate are anal swabs for detecting HSIL in this group?
* How does having HSIL affect the quality of life of MSM using PrEP?
* Can DNA methylation testing help improve our understanding of HSIL in these individuals?

Participants will:

* Answer questions about their health and quality of life.
* Have an anal smear collected for testing.
* Undergo High-Resolution Anoscopy (HRA) to check for HSIL and get a biopsy if deemed necessary.

DETAILED DESCRIPTION:
This study aims to evaluate High-Grade Squamous Intraepithelial Lesions (HSIL) in men who have sex with men (MSM) using Pre-Exposure Prophylaxis (PrEP) for HIV prevention. MSM are at increased risk for developing anal cancer, and HSIL is a known precursor to this type of cancer. The study seeks to assess the prevalence of HSIL, the screening accuracy of anal swabs, and the impact of HSIL on quality of life for MSM using PrEP. Furthermore, the study will explore the use of DNA methylation testing as a potential tool for improving the detection and understanding of HSIL in this high-risk group.

This multicenter clinical trial will involve MSM using PrEP at several study sites to ensure a diverse and representative sample.

The study will focus on prevalence, screening accuracy, and quality of life impacts, and will incorporate DNA methylation testing to explore potential molecular markers for early detection and progression of HSIL.

The primary goal of the study is to improve the early detection of HSIL in MSM using PrEP. By evaluating screening methods and quality of life, this study aims to provide valuable data that could lead to more effective screening strategies and interventions for preventing anal cancer in this population. The use of DNA methylation testing will provide additional insights into the molecular biology of HSIL, potentially informing future screening protocols.

This study addresses a significant gap in current research regarding the prevention and early detection of anal cancer in MSM using PrEP and aims to contribute critical data to improve healthcare outcomes for this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* HIV-uninfected MSM (men who have sex with men) aged 35 years or older.
* participants must have been using PrEP for at least 3 months.
* Dutch, English or French speaking and writing

Exclusion Criteria:

* Any intervention in the (peri-)anal region within the past 3 months
* Enema usage within 2 h before sampling
* Currently undergoing peri-anal topical HPV-treatment
* HRA in the last year (anal swab or HRA prior to the last year is no exclusion)

Min Age: 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of anal high-risk HPV infection in MSM-PrEP in Belgium | From screening to study completion for the patient (on average 8 months).
  The primary endpoint aims to determine the prevalence of HR HPV in MSM-PrEP in Belgium.

SECONDARY OUTCOMES:
Prevalence of abnormal anal cytology in MSM using PrEP in Belgium | From screening to study completion for the patient (on average 8 months).
  The secondary endpoint aims to determine the prevalence of abnormal anal cytology in MSM using PrEP in Belgium
Prevalence of abnormal histology, i.e. LSIL and HSIL in MSM using PrEP in Belgium | From screening to study completion for the patient (on average 8 months).
  The third endpoint aims to determine the prevalence of abnormal anal histology in MSM using PrEP in Belgium
Methylation on cytology (screening) samples and histology (HRA) samples | From screening to study completion for the patient (on average 8 months).
  The fourth endpoint aims to investigate methylation profiles according to the cytological or histo-logical results
Accuracy of anal HPV genotyping, anal cytology and methylation, together or as separate tests in the prediction of hHSIL | From screening to study completion for the patient (on average 8 months).
  The fifth endpoint aims to determinate the specificity and sensitivity of anal HPV genotyping, anal cytology and methylation, together and as separate tests, used as screening tests for hHSIL.
Can we distinguish different profiles in hHSIL suggesting repression or progression? | From screening to study completion for the patient (on average 8 months).
  profiling hHSIL in terms of methylation and biomarkers such as HPV genotyping, HPV-E4, p16 and Ki67
Can ASCL1/ZNF582 methylation test make accuracy of the less invasive anal swab testing better and/or be used to guide treatment decision making? | From screening to study completion for the patient (on average 8 months).
  Receiver operating curve analysis of anal swabs for hHSIL detection with or without methylation testing on anal swab.
Determine the incidence of HPV related lesions between demographics, lifestyle, HPV vaccination, sexual risk behavior, history of STI and HPV infection, cytology and histology. | From screening to study completion for the patient (on average 8 months).
  Determination of (multiple) correlations between demographics, lifestyle, HPV vaccination, sexual risk behavior, history of STIs versus HPV infection and abnormal cytohistology.
Impact of anal cancer screening in MSM using PrEP on quality of life | From screening to study completion for the patient (on average 8 months).
  Determination of quality of life using EQ-5D questionnaire (annex 1) at screening and follow-up in MSM using PrEP.

CONTACTS AND LOCATIONS:
Locations (7):
- Belgium (7):
  - AZ Sint Jan, Bruges
  - CHU Saint-Pierre, Brussels
  - Cliniques universitaires Saint-Luc - UCLouvain, Brussels
  - UZ Brussel, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - CHU Charleroi - Chimay, Lodelinsart

IPD SHARING:
Plan to Share IPD: Undecided